CLINICAL TRIAL: NCT01531244
Title: A Phase I/II Study of Isolated Limb Infusion and Targeted Gene Therapy for Advanced, Unresectable Extremity Melanoma
Brief Title: Isolated Limb Infusion Chemotherapy With Targeted Gene Therapy for Advanced, Unresectable Extremity Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-X335
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Dactinomycin; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (targeted gene therapy and ILI) (Experimental): Patients receive melphalan and dactinomycin via ILI. Patients then receive CRAd 3/5-delta via ILI.
  Interventions: Biological: dactinomycin; Drug: melphalan; Biological: Conditionally replicative adenovirus 3/5-delta

INTERVENTIONS:
Biological: dactinomycin — Given via ILI
  Other Names: ACT-D, actinomycin C1, actinomycin D, AD, Cosmegen, DACT
Drug: melphalan — Given via ILI
  Other Names: Alkeran, CB-3025, L-PAM, L-phenylalanine mustard, L-Sarcolysin, Melfalan
Biological: Conditionally replicative adenovirus 3/5-delta — Given via ILI
  Other Names: CRAd 3/5-delta

SUMMARY:
This phase I/II trial studies the safety, best dose and effectiveness of targeted gene therapy combined with isolated limb infusion (ILI) of melphalan and dactinomycin for treating patients with advanced extremity melanoma that cannot be removed by surgery. Adding gene therapy to a standard chemotherapy regimen in the isolated limb may enhance anti-cancer effects by inducing a systemic immune response against the tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed diagnosis of melanoma with advanced, unresectable primary or in transit metastasis
* Patient must have measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with caliper measurement for superficial lesions or computed tomography (CT) scan for deeper lesions; additionally, patients must have no evidence of disease beyond the affected extremity on positron emission tomography (PET)/CT scan
* Patients may have undergone any previous systemic chemotherapy with a treatment free period of > 4 weeks prior to enrolling on this clinical trial
* Patient must be > 18 years of age.-Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2, Karnofsky >= 60%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x IULN
* Creatinine within normal institutional limits
* OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately
* Patient (or legally authorized representative if applicable) must be able to understand and willing to sign an institutional review board (IRB) approved written informed consent document

Exclusion Criteria:

* Patients must not have had previous oncolytic viral therapy
* Patient must not be receiving any other investigational agents
* Patient must not have known brain metastases; patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to melphalan or dactinomycin or other agents used in the study
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient must not be pregnant and/or breastfeeding
* Patient must not be known to be human immunodeficiency virus (HIV)-positive or otherwise immunocompromised (i.e., patient has undergone organ/bone marrow transplant on immunosuppression, patient is or has recently undergone treatment with toxic chemotherapy for another malignancy, etc.) as there is a risk of complications in the use of adenovirus therapy in these patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Optimal tolerated dose (OTD) of CRAd 3/5 | 14 days
  Defined as the dose level at which > 50% of target lesion viral infectivity is achieved and < 2 of 6 patients have dose limiting toxicities.
Response rate (complete response [CR] + partial response [PR]) of CRAd 3/5-delta in combination with standard M-ILI (Phase II) | 3 months
  Assessed using revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Progression Free Survival (Phase II) | 2 years
  Duration of time from start of treatment to time of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Safety of CRAd 3/5-delta in combination with standard M-ILI | 2 years
  Descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Infectivity rate of CRAd 3/5-delta | 2 days; baseline and day 1 or 2 post treatment
  Lesion biopsies; quantified using immunohistochemical staining method.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Fields, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Background] Turley RS, Raymond AK, Tyler DS. Regional treatment strategies for in-transit melanoma metastasis. Surg Oncol Clin N Am. 2011 Jan;20(1):79-103. doi: 10.1016/j.soc.2010.09.008. PMID 21111960
- [Background] Aloia TA, Grubbs E, Onaitis M, Mosca PJ, Cheng TY, Seigler H, Tyler DS. Predictors of outcome after hyperthermic isolated limb perfusion: role of tumor response. Arch Surg. 2005 Nov;140(11):1115-20. doi: 10.1001/archsurg.140.11.1115. PMID 16301451
- [Background] Brady MS, Brown K, Patel A, Fisher C, Marx W. A phase II trial of isolated limb infusion with melphalan and dactinomycin for regional melanoma and soft tissue sarcoma of the extremity. Ann Surg Oncol. 2006 Aug;13(8):1123-9. doi: 10.1245/ASO.2006.05.003. Epub 2006 Jun 21. PMID 16791448
- [Background] Beasley GM, Riboh JC, Augustine CK, Zager JS, Hochwald SN, Grobmyer SR, Peterson B, Royal R, Ross MI, Tyler DS. Prospective multicenter phase II trial of systemic ADH-1 in combination with melphalan via isolated limb infusion in patients with advanced extremity melanoma. J Clin Oncol. 2011 Mar 20;29(9):1210-5. doi: 10.1200/JCO.2010.32.1224. Epub 2011 Feb 22. PMID 21343562
- [Background] Kroon HM, Moncrieff M, Kam PC, Thompson JF. Outcomes following isolated limb infusion for melanoma. A 14-year experience. Ann Surg Oncol. 2008 Nov;15(11):3003-13. doi: 10.1245/s10434-008-9954-6. Epub 2008 May 29. PMID 18509706
- [Background] Raymond AK, Beasley GM, Broadwater G, Augustine CK, Padussis JC, Turley R, Peterson B, Seigler H, Pruitt SK, Tyler DS. Current trends in regional therapy for melanoma: lessons learned from 225 regional chemotherapy treatments between 1995 and 2010 at a single institution. J Am Coll Surg. 2011 Aug;213(2):306-16. doi: 10.1016/j.jamcollsurg.2011.03.013. Epub 2011 Apr 13. PMID 21493111
- [Background] Alvarez RD, Barnes MN, Gomez-Navarro J, Wang M, Strong TV, Arafat W, Arani RB, Johnson MR, Roberts BL, Siegal GP, Curiel DT. A cancer gene therapy approach utilizing an anti-erbB-2 single-chain antibody-encoding adenovirus (AD21): a phase I trial. Clin Cancer Res. 2000 Aug;6(8):3081-7. PMID 10955787
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu